CLINICAL TRIAL: NCT03418662
Title: A Randomized Trial Comparing the Adenoma Detection Rates Between EndoRings Colonoscopy (EC) and Standard Colonoscopy (SC).
Brief Title: EndoRings Colonoscopy vs Standard Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: US Endoscopy (Industry)
Responsible Party: Principal Investigator, Douglas K. Rex, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1711224972
Record Dates: First submitted 2018-01-02; First posted 2018-02-01 (Actual); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Adenoma; Colorectal Polyp; Colon Cancer
Keywords: Colonoscopy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Arm (Standard Colonoscopy) (No Intervention): Standard colonoscopy with no device attachment.
- EndoRings Colonoscopy (Experimental): Colonoscopy with EndoRings device attached to the distal end of the scope.
  Interventions: Device: EndoRings device

INTERVENTIONS:
Device: EndoRings device — Subjects randomized to undergo a colonoscopy procedure with the EndoRings device will have the device placed on the colonoscope that will be used during their procedure.
  Arms: EndoRings Colonoscopy

SUMMARY:
The study aims to compare the results between a standard colonoscopy to a colonoscopy with an attachment on the distal end of the colonoscope.

DETAILED DESCRIPTION:
This will be a prospective, randomized controlled study. Subjects referred for screening or surveillance colonoscopy will be prospectively enrolled. This study aims to compare the adenoma detection rates between EndoRings colonoscopy (EC) and Standard colonoscopy (SC). It is assumed that the proportion of patients with at least one adenoma would be 25% with SC and 35% with EC.

ELIGIBILITY:
Inclusion Criteria:

* Screening or Surveillance Colonoscopy
* Able to provide written informed consent

Exclusion Criteria:

* Known narrow colon or colon stenosis
* Personal history of Colorectal cancer
* History of inflammatory bowel disease
* Familial adenomatous polyposis syndrome (FAP)
* Hyperplastic polyposis syndrome
* Referral for incomplete colonoscopy or polyp clearance

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Rex, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared upon the discretion of the principal investigator.

REFERENCES:
- [Derived] Rex DK, Kessler WR, Sagi SV, Rogers NA, Fischer M, Bohm ME, Wo JM, Dewitt JM, McHenry L, Lahr RE, Searight MP, MacPhail M, Sullivan AW, McWhinney CD, Vemulapalli KC. Impact of a ring-fitted cap on insertion time and adenoma detection: a randomized controlled trial. Gastrointest Endosc. 2020 Jan;91(1):115-120. doi: 10.1016/j.gie.2019.06.042. Epub 2019 Jul 9. PMID 31299257

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 592 patients were enrolled in the study, but 17 were excluded before randomization for not meeting inclusion criteria. 569 patients were randomized.
Period: Overall Study
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy)
Started | 287 | 282
Completed | 284 | 278
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy) | Total
Number analyzed (Participants) | 284 | 278 | 562
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (8.1) | 61.0 (7.9) | 61.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 142 | 273
  Male | 153 | 136 | 289
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 233 | 222 | 455
  Other | 51 | 56 | 107
Region of Enrollment [Number; unit: participants]
  United States | 284 | 278 | 562
Indication for Colonoscopy [Count of Participants; unit: Participants] — Colonoscopy in patients without previously discovered polyps and for no other reason than screening for colorectal cancer is termed Screening colonoscopy. If the patient had polyps in a prior colonoscopy, then the indication would be Surveillance colonoscopy.
  Participants
    Patients who had a screening colonoscopy | 143 | 162 | 305
    Patients who had a surveillance colonoscopy | 141 | 116 | 257

OUTCOME MEASURES:

1. Primary Outcome: Adenoma Detection Rates
Description: Number of participants with at least one adenoma detected, during Standard Colonoscopy compared with colonoscopy with EndoRings.
Time Frame: During colonoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy)
Number analyzed (Participants) | 284 | 278
Participants | 143 | 124

2. Primary Outcome: Number of Adenomas Per Colonoscopy
Description: Comparison of the number of adenomas detected per colonoscopy between standard colonoscopy and EndoRings colonoscopy.
Time Frame: During colonoscopy procedure
Measure: Mean (Standard Deviation); unit: adenomas per colonoscopy
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy)
Number analyzed (Participants) | 284 | 278
adenomas per colonoscopy | 1.46 (2.69) | 1.06 (1.83)

3. Secondary Outcome: Polyp Detection Rate
Description: Number of subjects with at least one polyp detected with Standard Colonoscopy compared to colonoscopy with EndoRings.
Time Frame: During colonoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy)
Number analyzed (Participants) | 284 | 278
Participants | 199 | 188

4. Secondary Outcome: Number of Detections Per Colonoscopy
Description: Comparison of the number of polyps detected per colonoscopy between EndoRings colonoscopy and Standard colonoscopy.
Time Frame: During colonoscopy procedure
Measure: Mean (Standard Deviation); unit: polyps per colonoscopy
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy)
Number analyzed (Participants) | 284 | 278
polyps per colonoscopy | 2.29 (3.09) | 1.82 (2.19)

5. Secondary Outcome: Total Number of Detections
Description: Comparison of the total number of polyps detected and the total number of adenomas detected between EndoRings colonoscopy and Standard colonoscopy.
Time Frame: During colonoscopy procedure
Measure: Number; unit: Detections
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy)
Number analyzed (Participants) | 284 | 278
Detections
  Polyps | 415 | 295
  Adenomas | 650 | 506

6. Secondary Outcome: Cecal Intubation Rate
Description: Comparison of cecal intubation rate (the number of procedures where the colonoscope was able to be inserted all the way to the cecum) between standard colonoscopy and EndoRings colonoscopy.
Time Frame: During colonoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy)
Number analyzed (Participants) | 284 | 278
Participants | 281 | 277

7. Secondary Outcome: Time Comparison for Each Method
Description: Comparison of the time required to reach the cecum, withdrawal time, and total procedure time.
  Insertion time: time required to reach the cecum Withdrawal time: time calculated from when withdrawing is started in the cecum till the colonoscope is removed. This includes time spent washing, inspecting the colon and removing polyps.
  Total procedure time: This is the sum of insertion and withdrawal times along with any time spent washing or removing polyps while in the cecum (before starting withdrawal).
Time Frame: During colonoscopy procedure
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy)
Number analyzed (Participants) | 284 | 278
Minutes
  Insertion Time | 6.3 (4.4) | 5.5 (3.4)
  Total Withdrawal Time | 11.8 (6.1) | 12.8 (5.9)
  Total Procedure Time | 19.4 (8.2) | 19.5 (7.9)

8. Secondary Outcome: Patient Comfort Score
Description: Comparison of patient comfort between Standard colonoscopy and EndoRings colonoscopy on a scale of 0 to 10 with 0 being no pain (best outcome) and 10 being worst imaginable pain (worst outcome).
Time Frame: After colonoscopy was completed while patient was in recovery area of endoscopy unit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy)
Number analyzed (Participants) | 284 | 278
units on a scale | 0.47 (1.1) | 0.36 (0.9)

9. Secondary Outcome: Problems Encountered With Equipment
Description: Occurrences of slippage of EndoRings or of device being removed on insertion.
Time Frame: During colonoscopy procedure
Population: This outcome measure is not applicable for patients randomized to the standard arm because there is no device attached in the standard arm of the study. For this reason, 0 patients are reported for the standard arm for this specific outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy)
Number analyzed (Participants) | 284 | 0
Participants
  Procedures with slippage of device | 17 |
  Procedures where device was removed | 25 |

ADVERSE EVENTS:
Time Frame: During the colonoscopy procedure and while the patient was in the recovery section of the endoscopy suite immediately after the procedure.
Arm/Group | EndoRings Colonoscopy | Control Arm (Standard Colonoscopy)
All-Cause Mortality (participants affected / at risk) | 0/284 | 0/278
Serious Adverse Events (participants affected / at risk) | 0/284 | 0/278
Other Adverse Events (participants affected / at risk) | 0/284 | 0/278

LIMITATIONS AND CAVEATS:
Single center design; Inability to blind endoscopists to device randomization; Most patients were sedated with propofol so it would not reasonably be expected to have a difference in patient comfort score

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT03418662/Prot_SAP_000.pdf